CLINICAL TRIAL: NCT06245213
Title: A Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Electrophysiology of ANAVEX3-71 in Adult Patients With Schizophrenia in a Multiple Ascending Dose Study (Part A), Followed by a Double-Blind, Randomized, Placebo-Controlled Study (Part B)
Brief Title: A Study of ANAVEX3-71 in Adults With Schizophrenia
Acronym: SZ-001
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Collaborators: COGNISION (Unknown); Cognitive Research Corporation (Industry); Hassman Research Institute (Unknown)
Responsible Party: Principal Investigator, Kathy Skoff, Investigator, Anavex Life Sciences Corp.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAVEX3-71-SZ-001
Record Dates: First submitted 2024-01-19; First posted 2024-02-07 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; EEG; Multiple Ascending Dose; Interventional; Sigma-1 Receptor Agonist; M1 Muscarinic Receptor Agonist; Biomarkers; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment in Part A and Part B. Part A: n = 16; Part B: n = 55;
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- ANAVEX3-71 30 mg TID (Part A) (Active Comparator): The first active treatment arm of the study during Part A (multiple ascending doses).
  Interventions: Drug: ANAVEX3-71 oral capsules
- ANAVEX3-71 60 mg TID (Part A) (Active Comparator): The second active treatment arm of the study during Part A (multiple ascending doses).
  Interventions: Drug: ANAVEX3-71 oral capsules
- ANAVEX3-71 Placebo TID (Part A) (Placebo Comparator): The placebo arm of Part A (multiple ascending doses).
  Interventions: Drug: Placebo oral capsules
- ANAVEX3-71 TBD mg TID (Part B) (Active Comparator): The active arm of Part B of the study. The dose will be determined based on data obtained in Part A.
  Interventions: Drug: ANAVEX3-71 oral capsules
- ANAVEX3-71 Placebo TID (Part B) (Placebo Comparator): The placebo arm of Part B of the study.
  Interventions: Drug: Placebo oral capsules

INTERVENTIONS:
Drug: ANAVEX3-71 oral capsules — ANAVEX®3-71 (formerly AF710B) is a dual SIGMAR1 receptor agonist and M1 positive allosteric modulator with agonistic effects. This novel mechanism of action offers the potential to treat all symptom domains (positive, negative, and cognitive) of schizophrenia without the side effects of standard of care antipsychotics.
  Arms: ANAVEX3-71 30 mg TID (Part A); ANAVEX3-71 60 mg TID (Part A); ANAVEX3-71 TBD mg TID (Part B)
Drug: Placebo oral capsules — The placebo comparator for the study.
  Arms: ANAVEX3-71 Placebo TID (Part A); ANAVEX3-71 Placebo TID (Part B)

SUMMARY:
A study to evaluate the safety, tolerability, efficacy, pharmacokinetics, and electrophysiology of ANAVEX3-71 in patients with Schizophrenia.

DETAILED DESCRIPTION:
ANAVEX3-71-SZ-001 is a two-part study. The first part is Part A: Multiple Ascending Dose, PK, safety, and dose selection. The second part is Part B: Double Blind, Placebo Controlled for exploratory efficacy and continued repeat-dose safety. This study will investigate the effects of ANAVEX3-71 in patients with Schizophrenia for the first time. This is an in-patient study. In both parts, participants will undergo either 10 or 28 days of dosing (Part A and Part B, respectively). Standard clinical outcome measures used in the clinic and novel fluid and electrophysiological biomarkers will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers 18-55 years of age, inclusive at screening.
2. Has a primary diagnosis of schizophrenia, for ≥ 1 year
3. Stable schizophrenia psychiatric symptoms for at least 6 weeks prior to screening.
4. Schizophrenia clinical symptom severity defined by meeting ALL of the following per the Positive and Negative Syndrome Scale (PANSS) item scores at screening:

   1. Delusions (P1) ≤ 4
   2. Hallucinatory behavior (P3) ≤ 4
   3. Unusual thought content (G9) ≤ 4
   4. Hostility (P7) ≤ 4
5. Patient has a PANSS total score ≤ 80 at screening and baseline visits and no worsening in PANSS total score between screening and baseline, of more than 20%.
6. Has a Brief Assessment of Cognition (BACS) T-score < 50 at the screening visit.
7. On a stable regimen of at least one and up to a maximum of two second-generation ("atypical") antipsychotic medications for at least 6 weeks prior to screening and agree to stay on this regimen for their entire study participation, with the following exceptions:

   1. Clozapine use is not permitted
   2. Quetiapine for sleep at doses less than 300 mg are permitted.
   3. Day time (including morning) quetiapine use as the background antipsychotic is not permitted.
8. Able to understand the requirements of the study and able and willing to provide written informed consent and to abide by the study procedures, in the judgment of the Investigator, including able and willing to remain in an in-patient setting during the study.
9. If of childbearing potential, using adequate contraceptive methods for the duration of the study.
10. Body mass index of 18.5 to 40.0 kg/m2 (inclusive) and total body weight > 50 kg (110 lbs.) for males and > 40 kg (88 lbs.) for females.
11. Has a negative urine screen for drugs of abuse and negative alcohol breath test at screening and check-in.
12. Patient resides in a stable living situation and is anticipated to return to that same stable living situation.

Exclusion Criteria:

1. Participation in a schizophrenia study in which the patient has received any investigational medications within 60 days prior to the baseline visit.
2. History or presence of a clinically significant, poorly treated, or unstable conditions that would jeopardize the safety of the patient or the validity of the study results.
3. Clinically significant abnormal findings on the physical examination, medical history, ECG, or clinical laboratory results at screening.
4. Calgary Depression Scale for schizophrenia (CDSS) score ≥6 at the screening or baseline visits.
5. Simpson Angus Scale (SAS) total score ≥5 at the screening and baseline visits at the screening or baseline visits.
6. Abnormal Involuntary Movement (AIMS) score of 2 for two or more movements or a score of 3 or 4 for any single movement on this scale at the screening or baseline visits.
7. Any primary the DSM-5-TR (American Psychiatric Association 2022) disorder other than schizophrenia within 12 months before screening (confirmed using MINI version 7.0.2 at screening).
8. Pregnant, lactating, or less than 3 months postpartum. Sperm donation is not allowed for 90 days after the final dose of study drug.
9. Risk for suicidal behavior during the study.
10. Inability to detect a 1000 Hz tone at 40 dB in both ears at screening.
11. Has psychiatric hospitalization(s) for more than 30 days (cumulative) during the 90 days before screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Single Dose Maximum Observed Plasma Concentration (Cmax) | Part A: Day 1
  Pharmacokinetic blood measurements of ANAVEX3-71 and metabolite M8 at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose.
Multiple Dose Maximum Observed Plasma Concentration (Cmax) | Part A: Day 1 and Day 9
  Pharmacokinetic blood measurements of ANAVEX3-71 and metabolite M8 at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose.
Cmax (steady state) | Part A: Day 1 and Day 9
  The maximum plasma concentration of ANAVEX3-71 and metabolite M8 after reaching a steady state. With measurements taken at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose on Days 1 and 9.
Tmax (steady state) | Part A: Day 1 and Day 9
  The time to maximum plasma concentration of ANAVEX3-71 and metabolite M8 after reaching a steady state. With measurements taken at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose on Days 1 and 9.
AUC (steady state) | Part A: Day 1 and Day 9
  The area under the curve of the plasma concentration of ANAVEX3-71 and metabolite M8 after reaching a steady state. With measurements taken at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose on Days 1 and 9.
AUC (single state) | Part A: Day 1 and Day 9
  The area under the curve of the plasma concentration of ANAVEX3-71 and metabolite M8 after a single day of dosing. With measurements taken at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose on Days 1 and 9.
CL/F (steady state) | Part A: Day 1 and Day 9
  The oral clearance of ANAVEX3-71 and metabolite M8 after reaching a steady state. With measurements taken at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose on Days 1 and 9.
Vz/F (steady state) | Part A: Day 1 and Day 9
  The volume of distribution based on the terminal elimination phase following administration ANAVEX3-71 and metabolite M8 after reaching a steady state. With measurements taken at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose on Days 1 and 9.
T1/2 (steady state) | Part A: Day 1 and Day 9
  The time to elimination of half the quantity of ANAVEX3-71 and metabolite M8 after reaching a steady state. With measurements taken at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose on Days 1 and 9.
Rac (steady state) | Part A: Day 1 and Day 9
  The observed accumulation rate of ANAVEX3-71 and metabolite M8 after reaching a steady state. With measurements taken at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose on Days 1 and 9.
Rac, Cmax (steady state) | Part A: Day 1 and Day 9
  The observed accumulation ratio for Cmax of ANAVEX3-71 and metabolite M8 after reaching a steady state. With measurements taken at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose on Days 1 and 9.
PTR (steady state) | Part A: Day 1 and Day 9
  The peak-to-trough ratio at steady state for ANAVEX3-71 and metabolite M8 after reaching a steady state. With measurements taken at pre-dose, 0.5, 1, 2-, 3-, 4-, and 8-hours post-dose on Days 1 and 9.
Adverse Events | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by the number of participants with treatment-related adverse events and the number of treatment-related adverse events, as assessed by CTCAE v4.0.
Vital Signs | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in vital signs including heart rate (beats per minute), blood pressure (mmHg), respiration rate (breaths per minute), and body temperature (degrees centigrade). These measurements will be reported together for the investigator to assess their clinical relevance and relation to potential treatment emergent adverse events.
12-lead ECG (RR interval) | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in the time elapsed between two successive R-waves of the QRS signal on the electrocardiogram (in seconds).
12-lead ECG (P wave) | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in the electrical depolarization of the atria of the heart (in milliseconds).
12-lead ECG (PR interval) | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in the conduction between the atria and ventricles (in milliseconds).
12-lead ECG (PR segment) | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in the portion of the ECG from the end of the P wave to the beginning of the QRS complex as measured by the electrocardiogram.
12-lead ECG (QRS complex) | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in ventricular depolarization as measured by the Q, R, and S waves on the electrocardiogram.
12-lead ECG (ST segment) | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in the interval between ventricular depolarization and repolarization as represented by the end of the S wave and beginning of the T wave on the electrocardiogram.
12-lead ECG (T wave) | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in ventricular repolarization (in milliseconds).
12-lead ECG (QT interval) | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in ventricular depolarization and repolarization as represented by the interval between the QRS complex to the end of the T wave.
Clinical Safety Labs - Renal Panel | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in clinical safety laboratory parameters including glucose, calcium, phosphorus, blood urea nitrogen, creatinine, sodium, potassium, chloride, and bicarbonate. These measurements will be combined to report whether clinical safety labs are abnormal and/or clinically significant by the investigator.
Clinical Safety Labs - Hepatic Panel | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in clinical safety laboratory parameters including albumin, alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, total bilirubin, direct bilirubin, indirect bilirubin, total protein, lactate dehydrogenase, and gamma-glutamyl transferase. These measurements will be combined to report whether clinical safety labs are abnormal and/or clinically significant by the investigator.
Clinical Safety Labs - Lipid Panel | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in clinical safety laboratory parameters including triglycerides, cholesterol (low-density lipoprotein [LDL], high-density lipoprotein [HDL]), and creatine phosphokinase.These measurements will be combined to report whether clinical safety labs are abnormal and/or clinically significant by the investigator.
Clinical Safety Labs - Hematology Panel | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in clinical safety laboratory parameters including Red blood cell (RBC) count, hemoglobin, hematocrit, white blood cell counts with differential, platelet count, RBC indices (mean corpuscular volume [MCV], mean corpuscular hemoglobin [MCH], and mean corpuscular hemoglobin concentration [MCHC]) and if RBC indices are abnormal, and reflex to RBC morphology if indices are abnormal.These measurements will be combined to report whether clinical safety labs are abnormal and/or clinically significant by the investigator.
Clinical Safety Labs - Urinalysis Panel | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in clinical safety laboratory parameters including Protein, glucose, pH, blood, leukocytes, leukocyte esterase, urobilinogen, bilirubin, ketones, and nitrite. These measurements will be combined to report whether clinical safety labs are abnormal and/or clinically significant by the investigator.
Clinical Safety Labs - Coagulation Panel | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in clinical safety laboratory parameters including activated partial thromboplastin time, prothrombin time, and international normalized ratio.These measurements will be combined to report whether clinical safety labs are abnormal and/or clinically significant by the investigator.
Brief Physical Examination | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in the general appearance of nails, skin, hair, body habitus, movement coordination, odors, breathing pattern, eyes, ears, nose, mouth, face, salivary glands, lymph nodes, thyroid, anterior and posterior torso, proximal/distal motor strength, and distal pulses. These measurements are combined to assess the general neurological status of the participant to report abnormalities and/or clinical significance by the investigator.
Brief Neurological Examination | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in the participant's mental status, gait, truncal stability, motor function, and visual capabilities. These measurements are combined to assess the general neurological status of the participant to report abnormalities and/or clinical significance by the investigator.
AIMS | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in the Abnormal Involuntary Movement Scale (AIMS). This is a rating scale that was designed to measure involuntary movements known as tardive dyskinesia (TD), which sometimes develops as a side effect of long-term treatment with neuroleptic (anti-psychotic) medications. The test, which can be completed in about 5 minutes, has a total of twelve items rating involuntary movements of various areas of the patient's body. Items are scored on a 0 (none) to 4 (severe) basis; the scale provides a total score (items 1 through 7) or item 8 can be used in isolation as an indication of overall severity of symptoms.
SAS | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  Safety as measured by changes in the Simpson-Angus Scale (SAS), administered typically within 5 minutes, it is a performance scale that measures anti-psychotic-induced parkinsonism symptoms. The rater asks the patient to perform 10 tasks and rates responses on a scale of 0-4 (normal to severe).
BARS | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  The Brief Adherence Rating Scale (BARS), administered typically within 5 minutes, is a 4-item questionnaire to assess a patient's adherence with their currently prescribed medication regimen. Medication non-adherence is common in patients with psychiatric conditions and associated with worse clinical outcomes. The BARS assesses a patient's compliance with their prescribed medication regimen. The tool is administered by a clinician and includes 4 items: 3 questions and an overall visual analog rating scale to estimate the proportion of doses taken by the patient in the past month (0-100%). The three questions probe patients' knowledge about their medication regimen: number of prescribed doses per day, number of days the patient did not take the prescribe dose, and number of days the patient took less than the prescribed dose.
CDSS | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  The Calgary Depression Scale for Schizophrenia (CDSS) is a 9-item clinician-rated outcome measure that assesses the level of depression in people with schizophrenia spectrum disorder, including attenuated psychosis syndrome. It distinguishes depressive symptoms from negative, positive, and extrapyramidal symptoms. The scales take approximately 10 minutes to administer and has a lookback period of 2-weeks. Each item is rated on a scale of 0-3 (absent to severe).
C-SSRS | Part A and Part B Screening to Safety Follow Up Visit; Up to 78 days (Part A) and Up to 114 days (Part B)
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a suicidal ideation rating scale. The scale identifies behaviors and thoughts that are associated with an increased risk of suicidal actions in the future. The C-SSRS baseline/screening version will be conducted at screening. The C-SSRS Since Last Visit version will be conducted for all visits after screening. Answers are "Yes" or "No" with the opportunity for the participant to explain their answers further.
EEG-ERP - Passive, Duration Deviant, Oddball ERP | Part A and Part B: Up to 12 days (Part A) and Up to 30 days (PartB)
  Electroencephalography (EEG) and event-related potential (ERP) measures of the duration deviant mismatch negativity paradigm. In this paradigm, 2 tones of the same frequency and sound intensity, one short duration (Standard) and one longer duration (Deviant), are sequentially presented to the patient through inserted earphones. Standard stimuli are presented more often than Deviant stimuli. While the auditory stimuli are being played, the patient is instructed to perform a picture-word matching task where they press a button on the COGNISON® handset when they see a picture and a word on a monitor positioned in front of them that do not match.
EEG-ERP - Active, Auditory, Oddball ERP | Part A and Part B: Up to 12 days (Part A) and Up to 30 days (PartB)
  Electroencephalography (EEG) and event-related potential (ERP) measures. In this paradigm, 2 tones of the same sound intensity, one low frequency (Standard) and one higher frequency (Target) are sequentially presented to the patient through inserted earphones. The Standard stimuli are presented more often than the Target stimuli. The patient is told to listen for the high-frequency stimuli (Target) and press a button on the COGNISION® handset as fast as they can.
EEG-ERP - Auditory Steady State Response | Part A and Part B: Up to 12 days (Part A) and Up to 30 days (PartB)
  Electroencephalography (EEG) and event-related potential (ERP) measures. In this paradigm, a short stream of clicks is repeatedly presented to the patient through inserted earphones. While the click-streams are being presented, the patient is instructed to fix their gaze on a white cross displayed on a computer monitor positioned in front of them.
EEG-ERP - Resting EEG | Part A and Part B: Up to 12 days (Part A) and Up to 30 days (PartB)
  Electroencephalography (EEG) and event-related potential (ERP) measures. In this paradigm, the patient is asked to close their eyes and relax for 5 minutes while EEGs are recorded.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Part A and Part B: Up to 12 days (Part A) and Up to 30 days (PartB)
  The Positive and Negative Syndrome Scale (PANSS) is an approximate 30-minute structured interview scale used for measuring the symptom severity of patients with schizophrenia. It is widely used in the study of antipsychotic therapy.
Brief Assessment of Cognition in Schizophrenia (BACS) | Part A and Part B: Up to 12 days (Part A) and Up to 30 days (PartB)
  The Brief Assessment of Cognition in Schizophrenia (BACS) assesses the aspects of cognition found to be most impaired and most strongly correlated with outcomes in patients with schizophrenia. The BACS requires less than 35 min to complete.
Clinical Global Impressions Scale Schizophrenia (CGI-SCH) | Part A and Part B: Up to 12 days (Part A) and Up to 30 days (PartB)
  The Clinical Global Impression-Schizophrenia Scale (CGI-SCH) assesses the positive, negative, depressive, cognitive symptoms, and overall severity of schizophrenia. The (CGI-SCH) scale is a brief assessment instrument which is originally adapted from the Clinical Global Impression (CGI) scale and the CGI Bipolar Patients (CGI-BP) scale. It was developed to study the outcome of antipsychotic treatment in schizophrenia in an observational study (Schizophrenia Outpatient Health Outcomes (SOHO) Study. The CGI-SCH has shown strong validity, and it has slightly higher interrater reliability than the PANSS (Kumari et al., 2017).
Virtual Reality Functional Capacity Assessment Tool (VRFCAT) | Part A and Part B: Up to 12 days (Part A) and Up to 30 days (PartB)
  The Virtual Reality Functional Capacity Assessment Tool (VRFCAT) is a computerized measure that was developed to be a reliable, valid, and sensitive measure of functional capacity, with the potential to demonstrate real-world functional improvements associated with cognitive change. The VRFCAT, typically administered within 15 minutes, presents patients with a realistic simulated environment to re-create routine activities of daily living, including, e.g., exploring a kitchen, catching a bus to a grocery store, finding/purchasing food in a grocery store, and returning home on a bus. To permit repeated testing while avoiding learning effects, 6 alternate forms were created that vary the ingredients stored in the cabinets, items on the recipe and grocery list, cost of the bus rides, cost of groceries, and money available in a wallet.
Blood measurements of chitinase-3-like protein 1 (YKL-40) | Part B: Baseline to End of Treatment (Day -2 to Day 28)
  Previous studies have identified genetic variants of the chitinase-3-like protein 1 gene (which expresses YKL-40) and elevated serum YKL-40 with an increased risk for schizophrenia in certain populations (Ohi et al., 2010). Subsequent studies in broader populations demonstrated monocyte activation and elevated YKL-40 in the plasma and cerebrospinal fluid of patients experiencing first-episode psychosis (Orhan et al., 2018). This study seeks to explore blood levels of YKL-40 before and after treatment with ANAVEX3-71 to investigate the immune calming effects associated with Sigma-1 receptor activation in patients with schizophrenia. The expected effect of Sigma-1 activation on inflammation may be an upstream effect by attenuating disease-related, chronic pro-inflammatory signaling by monocytes and glia, to prevent downstream injury due to inflammation (Zhang et al., 2023).
Blood measurements of glial fibrillary acidic protein (GFAP) | Part B: Baseline to End of Treatment (Day -2 to Day 28)
  Immune dysfunction theories of schizophrenia include glial-related dysfunction and assume that initial disturbances in glial cells can lead or contribute to neuronal abnormalities that drive symptoms of schizophrenia. Glial perturbations in schizophrenia are associated with a neuroinflammatory response and elevated levels of glial fibrillary acidic protein (GFAP) (Wang et al., 2015).
Blood measurements of circulating amino acid metabolites | Part B: Baseline to End of Treatment (Day -2 to Day 28)
  Changes in the metabolomic profile of circulating amino acids and related metabolites are implicated in the etiology of numerous neurological and neuropsychiatric disorders (Donatti et al., 2020). Metabolomics studies of patients with schizophrenia demonstrate numerous metabolite signatures of schizophrenia including elevated glutamate (Davison et al., 2018). Changes in these metabolite levels may result from treatment, based on previous research into the treatment of other central nervous system disorders with Sigma-1 receptor agonists such as ANAVEX3-71.
Exploratory DNA/RNA, including whole genome analysis and whole transcriptome mRNA | Part B: Baseline to End of Treatment (Day -2 to Day 28)
  Exploratory DNA/RNA, including whole genome analysis and whole transcriptome mRNA. Assessed in whole blood via next generation sequencing (NGS) method. Whole genome sequencing (WGS) with 30x read depth. These measurements will be used to understand the potential effects of genetic variation on treatment response and the potential effect of treatment on changes in gene expression which may be relevant to the etiology of schizophrenia.

CONTACTS AND LOCATIONS:
Locations (1):
- CenExel Hassman Research Institute, Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided